CLINICAL TRIAL: NCT06215118
Title: A PHASE 1B, OPEN-LABEL STUDY OF ELRANATAMAB IN COMBINATION WITH IBERDOMIDE IN PARTICIPANTS WITH RELAPSED REFRACTORY MULTIPLE MYELOMA
Brief Title: A Study to Learn About the Effects of the Combination of Elranatamab (PF-06863135) and Iberdomide in Patients With Relapsed or Refractory Multiple Myeloma (MagnetisMM-30)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C1071030; MagnetisMM-30 (Other: Alias Study Number)
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
Keywords: elranatamab; PF-06863135; iberdomide; relapsed; refractory; RRMM; BCMA; MagnetisMM; Bispecific antibody; CC-220
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Dose Escalation (Experimental): Non-randomized elranatamab plus iberdomide
  Interventions: Drug: Elranatamab; Drug: Iberdomide
- Part 2 Dose Randomization (Experimental): Randomized elranatamab plus iberdomide
  Interventions: Drug: Elranatamab; Drug: Iberdomide

INTERVENTIONS:
Drug: Elranatamab — BCMA-CD3 bispecific antibody
  Other Names: PF-06863135
Drug: Iberdomide — cereblon-modulating agent
  Other Names: CC-220; BMS-986382

SUMMARY:
The main purpose of the study is to understand how safe and tolerable is elranatamab when given along with iberdomide.

There are 2 parts to this study. Part 1 will look at how safe and tolerable is elranatamab when given with iberdomide. Part 2 will look at the correct amount of this combination that can be given to patients with relapsed or refractory multiple myeloma.

Myeloma is a type of cancer that begins in plasma cells (white blood cells that produce antibodies). Refractory means a disease or condition that does not respond to treatment. Relapsed means the return of a disease after a period of improvement.

All study medicines are given in cycles that last 28 days. Everyone taking part in this study will receive elranatamab as a shot under the skin. Iberdomide will be taken by mouth once a day for 21 days over a 28-day cycle.

Participants will receive study medicine until:

* their disease progresses or,
* they experience unacceptable side effects or,
* they choose to no longer take part in the study.

The study will look at the experiences of people receiving the study medicines. This will help see if the study medicines are safe and can be used for multiple myeloma treatment.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of multiple myeloma as defined by IMWG criteria
* Measurable disease based on IMWG criteria as defined by at least 1 of the following:
* Serum M-protein ≥0.5 g/dL by SPEP
* Urinary M-protein excretion ≥200 mg/24 hour by UPEP
* Serum immunoglobulin FLC ≥10 mg/dL (≥100 mg/L) AND abnormal serum immunoglobulin kappa to lambda FL ratio (<0.26 or >1.65)
* Part 1: Received 2-4 prior lines of therapy for multiple myeloma, consisting of at least 1 immunomodulatory drug and 1 proteasome inhibitor.
* Part 2: Received 1-3 prior lines of therapy for multiple myeloma, consisting of at least 1 immunomodulatory drug and 1 proteasome inhibitor.
* ECOG performance status 0-1
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1

Exclusion Criteria:

* Plasma cell leukemia, Smoldering multiple myeloma, Waldenström's macroglobulinemia, Amyloidosis, POEMS Syndrome
* Impaired cardiovascular function or clinically significant cardiovascular diseases
* Stem cell transplant within 12 weeks prior to enrollment or active graft vs host disease
* Participants with any active, uncontrolled bacterial, fungal, or viral infection
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ
* Previous treatment with:
* BCMA-directed or CD3 redirecting therapy
* Iberdomide (CC-220) or Mezigdomide
* Administration of strong inhibitor or inducer of CYP3A4/5 within 2 weeks prior to dosing and during the study
* Administration with an investigational product within 30 days preceding the first dose of study intervention
* Participant is unable or unwilling to undergo protocol required thromboembolism prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2027-04-10 (Estimated); Study Completion 2028-03-09 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with dose limiting toxicity (DLT) | Cycle 1, about 28 days
  Dose limiting toxicity rate based on dose limiting toxicity evaluable participants
Part 2: Number of participants with Adverse Events (AE) by Seriousness and Relationship to Treatment | Assessed from baseline up to 90 days after last dose of study treatment
  Number of participants with AE among participants who take at least 1 dose of study intervention. AEs are categorized by seriousness and relationship to treatment. Relatedness to study drug is assessed by investigator.

SECONDARY OUTCOMES:
Part 1: Number of participants with Adverse Events (AE) by Seriousness and Relationship to Treatment | Assessed from baseline up to 90 days after last dose of study treatment
  Number of participants with AE among participants who take at least 1 dose of study intervention. AEs are categorized by seriousness and relationship to treatment. Relatedness to study drug is assessed by investigator.
Part 1 and Part 2: Number of Participants with Adverse Events (AE) characterized by type, frequency, severity | Assessed from baseline up to 90 days after last dose of study treatment
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibly of causal relationship
Part 1 and Part 2: Number of Participants with Clinically Significant Change from Baseline in Laboratory Abnormalities | Assessed from baseline up to 90 days after last dose of study treatment
  Laboratory abnormalities as characterized by type, frequency, severity
Part 1 and Part 2: Percentage of Participants with Objective Response Rate (ORR) | Assessed for approximately 2 years
  Percent of participants having confirmed Stringent Complete Response (sCR), Complete Response (CR), Very Good Partial Response (VGPR), or Partial Response (PR) per IMWG criteria as determined by investigator
Part 1 and Part 2: Percentage of Participants with Complete Response Rate (CRR) | Assessed for approximately 2 years
  Percent of participants having Complete Response/ Stringent Complete Response (CR+sCR) per IMWG criteria as determined by investigator
Part 1 and Part 2: Time to Response (TTR) | Assessed for approximately 2 years
  For participants with an objective response per IMWG criteria, TTR is the time from first dose to the first documentation of objective response that is subsequently confirmed
Part 1 and Part 2: Duration of Response (DOR) | Assessed for approximately 2 years
  For participants with an objective response per IMWG criteria, DOR is the time from first documentation of objective response that is subsequently confirmed until the first documentation of confirmed progressive disease (PD) per IMWG criteria
Part 1 and Part 2: Duration of Complete Response (DOCR) | Assessed for approximately 2 years
  For participants with a Complete Response/ Stringent Complete Response (CR+sCR) per IMWG criteria, DOCR is the time from the first documentation of CR/sCR that is subsequently confirmed until the first documentation of confirmed progressive disease (PD) per IMWG criteria
Part 1 and Part 2: Time of Progression Free Survival (PFS) | Assessed for approximately 2 years
  Progression free survival (IMWG criteria)
Part 1 and Part 2: Time of Overall Survival (OS) | Assessed for approximately 2 years
  The duration of time from first dose of study treatment to death
Part 1 and Part 2: Minimal Residual Disease (MRD) Negativity Rate | Assessed for approximately 2 years
  The proportion of participants achieving CR+sCR with negative MRD per IMWG sequencing criteria, from the date of first dose until the first documentation of confirmed progressive disease (PD), death, or start of new anticancer therapy.
Part 1 and Part 2: Concentrations of elranatamab | Assessed for approximately 2 years
  Pre-dose and post-dose concentrations of elranatamab
Part 1 and Part 2: Concentrations of iberdomide | Assessed for approximately 4 months
  Pre-dose concentrations of iberdomide
Part 1 and Part 2: Percentage of participants with positive anti-drug antibodies (ADA) against elranatamab | Assessed for approximately 2 years
  Percent of participants with positive ADA to elranatamab when given in combination with iberdomide

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (28):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Indiana CTSI Clinical Research Center (ICRC), Indianapolis, Indiana
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center (IUSCCC), Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Methodist Hospital, Omaha, Nebraska
  - Oncology Hematology West P.C. dba Nebraska Cancer - Methodist, Omaha, Nebraska
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack, Commack, New York
  - MSK Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center - Investigational Drug Service Pharmacy, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - MSK Nassau, Uniondale, New York
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Townsville University Hospital, Douglas, Queensland
  - Epworth Freemasons, East Melbourne, Victoria
  - Epworth Hospital, Richmond, Victoria
  - Slade Pharmacy, Richmond, Victoria
- Canada (3):
  - Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Univer, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071030